CLINICAL TRIAL: NCT05374928
Title: Human Epilepsy Project 3: Newly Diagnosed Idiopathic Generalized Epilepsy
Brief Title: Human Epilepsy Project 3
Acronym: HEP3
Status: Active, not recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 19-01030
Record Dates: First submitted 2022-05-11; First posted 2022-05-16 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Generalized Epilepsy
MeSH Terms: conditions — Epilepsy, Idiopathic Generalized

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will be asked to provide urine for small molecule analysis, blood if he/she is 13-17 years old, or protein, cell-free DNA, metabolomics, and RNA analyses, and a stool sample for microbiome analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Newly Diagnosed Idiopathic Generalized Epilepsy (IGE): Cohort 1 will have IGE that was diagnosed within the prior year. We will follow these participants for a minimum of two years.
- Cohort 2: Longstanding Treatment Responsive: Cohort 2 will consist of subjects with established IGE who have been responsive to treatment.
- Cohort 3: Longstanding IGE, Treatment Resistant: Cohort 3 will consist of patients with established treatment-resistant IGE.

SUMMARY:
By carrying a careful, large-scale and ambitious prospective study of a cohort of participants with generalized epilepsy, the study team hopes to clarify the likelihood of response and remission in this type of epilepsy, and try to explore the underlying biological drivers of treatment response, including novel realms of exploration such as impact of the microbiome, and genetics. The identification of biomarkers that predict the likelihood of disease response would allow epilepsy patients to make more informed decisions about the factors affecting their quality of life, including plans for driving, relationships, pregnancy, schooling, work, and play. In addition to its impact on clinical care, the data and specimens collected in HEP3, including sequential electrophysiology, biochemical profiles and neuroimaging and banked DNA for future genomics studies, have the potential to provide new insights into the biological basis of IGE, thereby advancing the discovery of effective treatments and cures. By enrolling both newly diagnosed subjects (prognosis unknown) as well as subjects with established IGE who are already determined to be treatment resistant or treatment responsive, the study team can immediately test potential biomarkers in a confirmation cohort, which will accelerate identification of predictive biomarkers.

ELIGIBILITY:
Cohort 1: Newly Diagnosed IGE

Inclusion criteria:

1. Age ≥13 years at time of enrollment
2. Age ≥8 years at time of seizure onset
3. Clinical seizure(s) and history consistent with IGE. The only permitted seizure types are absence, myoclonus or generalized tonic-clonic convulsions
4. Occurrence of at least 1 seizure of any type in the 6 months prior to treatment
5. Patients must have one of the following:

   * GTCSs alone accompanied by generalized spike-wave consistent with IGE per adjudication review
   * GTCSs with a history of absence and/or myoclonus, accompanied by generalized spike-wave consistent with IGE per adjudication review
   * GTCSs associated with a history of absence and/or myoclonus, not accompanied by generalized spike-wave consistent with IGE per adjudication review
   * A clear history of absence and/or myoclonus, accompanied by generalized spike-wave consistent with IGE per adjudication review
6. Availability of a complete medication history since initiation of treatment, including doses and date of initiation
7. No competing cause of epilepsy (e.g. traumatic brain injury)
8. AED treatment (for seizures) instituted not more than 12 months before enrollment

Exclusion Criteria

1. Focal epilepsy
2. Generalized/focal epilepsy mixed syndromes
3. Progressive neurological disorder (brain tumor, Alzheimer's disease, progressive myoclonic epilepsy, etc.)
4. Epileptic or developmental encephalopathy
5. Major medical co-morbidities (e.g. renal failure requiring dialysis, metastatic cancer, HIV, or significant liver or renal disease)
6. Autism Spectrum Disorder
7. History of chronic drug or alcohol abuse (misuse or excessive use that interferes with activities of daily living) within the last 2 years
8. Seizures only during pregnancy
9. History of previous or current significant psychiatric disorder that would interfere with study requirements

Cohort 2: Longstanding Treatment Responsive

Inclusion Criteria:

1. Age ≥13 years at time of enrollment
2. Age ≥8 years at time of seizure onset
3. Clinical seizure(s) and history consistent with IGE. The only permitted seizure types are absence, myoclonus or generalized tonic-clonic convulsions
4. Patients must have had one of the following:

   1. GTCSs alone accompanied by generalized spike-wave consistent with IGE per adjudication review
   2. GTCSs with a history of absence and/or myoclonus, accompanied by generalized spike-wave consistent with IGE per adjudication review
   3. GTCSs associated with a history of absence and/or myoclonus, not accompanied by generalized spike-wave consistent with IGE per adjudication review
   4. A clear history of absence and/or myoclonus, accompanied by generalized spike-wave consistent with IGE per adjudication review
5. Availability of a complete medication history since initiation of treatment, including doses and date of initiation
6. No competing cause of epilepsy (e.g. traumatic brain injury)
7. Two years of well-controlled seizures.

   1. No convulsive seizures in the last two years
   2. Myoclonic or absence seizures must be rare (<2 per year) and non-disabling
   3. Ongoing therapy with > 1 antiseizure medication

Exclusion Criteria:

1. Focal epilepsy
2. Paroxysmal nonepileptic seizures
3. Generalized/focal epilepsy mixed syndromes
4. Progressive neurological disorder (brain tumor, Alzheimer's disease, progressive myoclonic epilepsy, etc.)
5. Epileptic or developmental encephalopathy
6. Major medical co-morbidities (e.g. renal failure requiring dialysis, metastatic cancer, HIV, or significant liver or renal disease)
7. Autism Spectrum Disorder
8. History of chronic drug or alcohol abuse (misuse or excessive use that interferes with activities of daily living) within the last 2 years
9. Seizures only during pregnancy
10. History of previous or current significant psychiatric disorder that would interfere with study requirements

Cohort 3: Longstanding IGE, Treatment Resistant

Inclusion Criteria:

1. Age ≥13 years at time of enrollment
2. Age ≥8 years at time of seizure onset
3. Clinical seizure(s) and history consistent with IGE. The only permitted seizure types are absence, myoclonus or generalized tonic-clonic convulsions
4. Occurrence of at least 1 seizure of any type in the 6 months prior to treatment onset
5. Patients must have had one of the following:

   1. GTCSs alone accompanied by generalized spike-wave consistent with IGE per adjudication review
   2. GTCSs with a history of absence and/or myoclonus, accompanied by generalized spike-wave consistent with IGE per adjudication review
   3. GTCSs associated with a history of absence and/or myoclonus, not accompanied by generalized spike-wave consistent with IGE per adjudication review
   4. A clear history of absence and/or myoclonus, accompanied by generalized spike-wave consistent with IGE per adjudication review
6. Availability of a complete medication history since initiation of treatment. This should include doses and date of initiation if possible, but minimum information would include name of drug, approximate duration of administration and reason for discontinuation, if applicable.
7. No competing cause of epilepsy (e.g. traumatic brain injury)
8. Treatment resistant IGE

   1. Initiation of treatment at least 2 years prior to enrollment
   2. Treatment resistance, as defined by failure of adequate trials of two tolerated and appropriately chosen and used AED schedules (whether as monotherapies or in combination to achieve seizure freedom). ASMs taken at enrollment would count towards this minimum.
   3. Either or both of the following two:

   i. One GTCC per year over the last 2 years. ii. Any type of seizure at least every 3 months which can consist of either: disabling myoclonus or absence (in the opinion of the subject and investigator) or GTCC d. Such seizures were not primarily due to significant illness (e.g, URI is not significant unless temperature >101oF (38.3oC), nonadherence to antiseizure medications or >2 alcoholic beverages within 48 hrs of seizure e. Ongoing therapy with > 1 antiseizure medication

Exclusion Criteria:

1. Focal epilepsy
2. Paroxysmal nonepileptic seizures
3. Generalized/focal epilepsy mixed syndromes
4. Progressive neurological disorder (brain tumor, Alzheimer's disease, progressive myoclonic epilepsy, etc.)
5. Epileptic or developmental encephalopathy
6. Major medical co-morbidities (e.g. renal failure requiring dialysis, metastatic cancer, HIV, or significant liver or renal disease)
7. Autism Spectrum Disorder
8. History of chronic drug or alcohol abuse (misuse or excessive use that interferes with activities of daily living) within the last 2 years
9. Seizures only during pregnancy
10. History of previous or current significant psychiatric disorder that would interfere with study requirements
11. History of/suspicion of provoked seizures accounting for 25% or more of seizures over the prior 2 years (eg alcohol, non-adherence, significant sleep deprivation).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed IGE, as well as a cohort of subjects with established IGE.
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Individual Seizures | Baseline
  Self-reported via the Seer Seizure Diary App (https://app.seermedical.com)
Number of Cluster Seizures | Baseline
  Self-reported via the Seer Seizure Diary App (https://app.seermedical.com)
Number of episodes of non-adherence | Baseline
  Self-reported via the Seer Seizure Diary App (https://app.seermedical.com)
Average daily steps | Baseline
  Participants will be provided a Fitbit Inspire HR watch and will be trained to open an account on fitbit.com and synchronize their Fitbit watch data into their Fitbit cloud account. Daily steps is synchronized and collected for this study.
Average distance walked | Baseline
  Participants will be provided a Fitbit Inspire HR watch and will be trained to open an account on fitbit.com and synchronize their Fitbit watch data into their Fitbit cloud account. Daily steps is synchronized and collected for this study.
Average heart rate | Baseline
  Participants will be provided a Fitbit Inspire HR watch and will be trained to open an account on fitbit.com and synchronize their Fitbit watch data into their Fitbit cloud account. Daily steps is synchronized and collected for this study.
Average daily sleep duration | Baseline
  Participants will be provided a Fitbit Inspire HR watch and will be trained to open an account on fitbit.com and synchronize their Fitbit watch data into their Fitbit cloud account. Daily steps is synchronized and collected for this study. Using the Embleema Patient Web App, participants will be able to consult their activity and sleep data in interactive graphs.
Average daily wake duration | Baseline
  Participants will be provided a Fitbit Inspire HR watch and will be trained to open an account on fitbit.com and synchronize their Fitbit watch data into their Fitbit cloud account. Daily steps is synchronized and collected for this study. Using the Embleema Patient Web App, participants will be able to consult their activity and sleep data in interactive graphs.
Change in Quality of Life in Epilepsy Inventory-10 (QOLIE-10) Score | Baseline, Month 12
  QOLIE-10 assesses the patient's quality of life. There are 11 total items. The total score range is 10-51; with higher scores indicating greater impairment. The total score is the sum of scores for all questions divided by the number of items answered. Thus, if a patient skipped an item, it is not reflected in the total score.
Change in Quality of Life in Epilepsy Inventory-10 (QOLIE-10) Score | Baseline, Month 24
  QOLIE-10 assesses the patient's quality of life. There are 11 total items. The total score range is 10-51; with higher scores indicating greater impairment. The total score is the sum of scores for all questions divided by the number of items answered. Thus, if a patient skipped an item, it is not reflected in the total score.
Change in Quality of Life in Epilepsy Inventory-10 (QOLIE-10) Score | Month 12, Month 24
  QOLIE-10 assesses the patient's quality of life. There are 11 total items. The total score range is 10-51; with higher scores indicating greater impairment. The total score is the sum of scores for all questions divided by the number of items answered. Thus, if a patient skipped an item, it is not reflected in the total score.
Change in General Anxiety Disorder-7 Screener (GAD-7) Score | Baseline, Month 12
  This will only be reported for adults. GAD-7 consists of 7 problems. Participants report how often they have been bothered by the 7 problems over the last 2 weeks on a Likert Scale from 0 (not at all) to 3 (nearly every day). The total score range is 0-21; the higher the score, the more severe the anxiety. 0-4=minimal anxiety, 5-9=mild, 10-14=moderate, 15-21=severe anxiety.
Change in General Anxiety Disorder-7 Screener (GAD-7) Score | Baseline, Month 24
  This will only be reported for adults. GAD-7 consists of 7 problems. Participants report how often they have been bothered by the 7 problems over the last 2 weeks on a Likert Scale from 0 (not at all) to 3 (nearly every day). The total score range is 0-21; the higher the score, the more severe the anxiety. 0-4=minimal anxiety, 5-9=mild, 10-14=moderate, 15-21=severe anxiety.
Change in General Anxiety Disorder-7 Screener (GAD-7) Score | Month 12, Month 24
  This will only be reported for adults. GAD-7 consists of 7 problems. Participants report how often they have been bothered by the 7 problems over the last 2 weeks on a Likert Scale from 0 (not at all) to 3 (nearly every day). The total score range is 0-21; the higher the score, the more severe the anxiety. 0-4=minimal anxiety, 5-9=mild, 10-14=moderate, 15-21=severe anxiety.
Columbia Suicide Severity Rating Scale (C-SSRS) Score | Baseline
  C-SSRS systematically tracks suicidal ideation and behavior. The total score range is 0 (no ideation is present) - 5 (active suicidal ideation with specific plan and intent). The higher the score, the greater one's suicidal ideation. Any score greater than 0 is important and may indicate the need for mental health intervention
Columbia Suicide Severity Rating Scale (C-SSRS) Score | Month 12
  C-SSRS systematically tracks suicidal ideation and behavior. The total score range is 0 (no ideation is present) - 5 (active suicidal ideation with specific plan and intent). The higher the score, the greater one's suicidal ideation. Any score greater than 0 is important and may indicate the need for mental health intervention
Columbia Suicide Severity Rating Scale (C-SSRS) Score | Month 24
  C-SSRS systematically tracks suicidal ideation and behavior. The total score range is 0 (no ideation is present) - 5 (active suicidal ideation with specific plan and intent). The higher the score, the greater one's suicidal ideation. Any score greater than 0 is important and may indicate the need for mental health intervention
Cogstate Neuropsychological Assessment Score | Baseline
  The Cogstate is a battery of online computerized tests that assesses functions such as attention, memory, and processing speed. Scores are normalized to the range of 0-100th percentile based on speed of test completion and task accuracy. A higher percentile score indicates higher levels of cognitive functioning within the tested domain as compared to controls.
Cogstate Neuropsychological Assessment Score | Month 12
  The Cogstate is a battery of online computerized tests that assesses functions such as attention, memory, and processing speed. Scores are normalized to the range of 0-100th percentile based on speed of test completion and task accuracy. A higher percentile score indicates higher levels of cognitive functioning within the tested domain as compared to controls.
Cogstate Neuropsychological Assessment Score | Month 24
  The Cogstate is a battery of online computerized tests that assesses functions such as attention, memory, and processing speed. Scores are normalized to the range of 0-100th percentile based on speed of test completion and task accuracy. A higher percentile score indicates higher levels of cognitive functioning within the tested domain as compared to controls.
Wide Range Achievement Test (WRAT-4) Score | Baseline
  WRAT4 is an academic skills assessment which measures reading skills, math skills, spelling, and comprehension. Only the Word Reading portion of the assessment will be administered. The total raw score range is from 0-70, with a normalized score range of 55-145. The higher the score, the more advanced the participant's reading comprehension skills for their age range.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (17):
  - University of California San Francisco (UCSF), San Francisco, California
  - Yale University, New Haven, Connecticut
  - Georgetown University, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Maine Medical Center, Portland, Maine
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - Mid-Atlantic Epilepsy Sleep Center, Bethesda, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota Epilepsy Group, Saint Paul, Minnesota
  - Washington University, St Louis, Missouri
  - St. Barnabas Medical Center, Livingston, New Jersey
  - NYU Langone Health - Comprehensive Epilepsy Center (CEC), New York, New York
  - Mount Sinai Hospital, New York, New York
  - Northwell Health, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah Hospital, Salt Lake City, Utah
- Monash University, Melbourne, Clayton VIC, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Researchers who provide a methodologically sound proposal will have access to the data upon reasonable request. All requests for study data will be submitted using a standardized form that will be available on the HEP3 website (www.humanepilepsyproject.org).